CLINICAL TRIAL: NCT04901572
Title: Feasibility Clinical Study for Testing Performance and Usability of Q300 Device (QART Sperm Morphology) vs. Reference Staining Methods in Laboratory Environment Simulating Pre-ICSI Sperm Imaging of Live Sperm Cells.
Brief Title: Testing Performance and Usability of Q300 Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: QART Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: QISI-01
Record Dates: First submitted 2021-05-19; First posted 2021-05-25 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Up to 75 sperm samples will be evaluated using the Q300 system and a standard staining method for device feasibility testing. No other groups will be present in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QART Imaging (Other): Cells will be individually selected with the system's micromanipulator under bright-field imaging. The cells will be representative of the cell population to be selected in ICSI procedures, covering the entire range of human sperm cell dimensions. Each selected cell will be simultaneously imaged by the QART system in two modalities:
  1. Standard brightfield.
  2. QART's imaging methodology.
  Interventions: Diagnostic Test: QISI device

INTERVENTIONS:
Diagnostic Test: QISI device — QISI device will simulate its use in ICSI procedures and evaluate sperm cells according to WHO guidelines.

SUMMARY:
A data collection clinical study performed on live human spermatozoa samples. Spermatozoa are imaged by QART Q300TM microscopy system. For the feasibility 1st phase of the study, up to 75 donors are expected to participate. Study group will include sperm samples donated by the clinic's patients (recruited by the investigators from the clinic's patient database) and/or by healthy volunteers (responding to advertisement).

DETAILED DESCRIPTION:
Cells will be individually selected by the system, and will be representative of the cell population to be selected in ICSI procedures. Each selected cell will be imaged by the QART system and independently and blindly reviewed by an Embryologist(s) team. According to these, each cell will be scored as 'Normal' or 'Abnormal' per WHO guidelines. Sperm cells that were successfully imaged with Q300, will be individually stained. Each stained cell will be imaged by BFM and the non-labeled image will be digitally stored (BFM-NL). The BFM-NL Image will be independently and blindly reviewed by an Embryologist team and scored as 'Normal' or 'Abnormal' per their best discretion.

The database generated in this study will be used for (i) testing the performance accuracy of the Q300 system for sperm cell dimensional measurements, (ii) providing feedback to the study sponsor (QART Medical Ltd.) regarding the usability of the Q300 system, (iii) further improving and testing the accuracy of the QART Feature Extraction algorithms and (v) assisting in determining the inclusion/exclusion criteria for subsequent clinical stages. In final validation stages, the conventional staining results will be statistically compared with the Q300 feature extraction results for each individual sperm cell. During the study, ICSI laboratory personnel (at least 10) will evaluate the suggested use scenarios of the device; device components and user interface, the simplicity of use, duration of use, level of expertise required from the Q300 operator, clarity in the use sequences, and perceived added complexity compared with contemporary ICSI routine.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers
2. Patients recruited from the hospital's andrology/IVF departments
3. Male, Age >18
4. Patient signed on informed consent

Exclusion Criteria:

1. Severe Oligozoospermia (less than 1 million sperm cells after preparation).
2. Documented presence of infectious disease transmitted in sperm fluids (e.g. HIV, HBV, HCV, Covid-19)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 75 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate agreement between the Q300 results to the reference method | 1 Day
  Demonstrate agreement between Q300 results, and Chemically stained image. the Q300 results will be provided automatically for each individual cell that will be images by the system, the reference method measurements will be provided by core lab embryologist and using a marking tool application.
evaluate the repeatability of the Q300 device results and compare it to the reference method repeatability. | 1 Day
  repeatability of bot the device measurements and the reference method will be evaluated and compared.
agreement of individual sperm cell's classification will be compared between the Q300 device and the reference method. | 1 Day
  agreement of individual sperm cell's classification (comply with WHO2021 criteria or non comply) will be compared between the Q300 device automatic results and the reference method results.

SECONDARY OUTCOMES:
Usability of the Q300 device will be evaluated | 1 Day
  Usability of the Q300 device will be evaluated using usability questionnaire.

CONTACTS AND LOCATIONS:
Locations (4):
- Israel (4):
  - Barzilai Medical Center, Ashkelon
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No